CLINICAL TRIAL: NCT04279886
Title: Three-dimensional Scanning of the Chest: a Comparison Between Three Different Imaging Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-6130
Record Dates: First submitted 2020-01-14; First posted 2020-02-21 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-02

CONDITIONS: Chest Wall Disorder

STUDY DESIGN:
Intervention Model Description: All included healthy volunteers received 6 three-dimensional scans, utilizing 3 different scanning systems (2 scans per system)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three-dimensional scan arm (Other)
  Interventions: Other: Three-dimensional scans

INTERVENTIONS:
Other: Three-dimensional scans — All included healthy volunteers received 6 three-dimensional scans, utilizing 3 different scanning systems (2 scans per system)

SUMMARY:
Recently, three-dimensional scanning of the torso has been proposed as an alternative for two-view chest radiographies and computed tomography to determine the severity of pectus excavatum without exposure to ionizing radiation. The range of three-dimensional scanning systems is broad with even varying systems being used within hospitals. Most of these scanning systems have been validated for accuracy and reproducibility, no comparison between these systems is known. In addition, severity measures of pectus excavatum, as well as other research outcomes, surgical planning techniques, and analysis methods are based on a single imaging system. It is subsequently essential to determine whether different imaging systems can be used interchangeably regarding accuracy and reproducibility.

The aim of this study was to assess the reproducibility and accuracy between three commonly used three-dimensional scanning systems.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers only

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Reproducibility | 1 month
  Mean difference between subsequent scans utilizing the same three-dimensional scanning system
Accuracy | 1 month
  Mean difference between scans, acquired by different three-dimensional scanning systems

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Centre, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided